CLINICAL TRIAL: NCT00779519
Title: A Prospective, Double-Blind, Randomized, Placebo-Controlled, Phase IIa, Multiple Dose, Multicenter Study to Assess Safety and Tolerability of TTP435 in Obese (Class 1-2) Subjects Over 8 Weeks of Treatment
Brief Title: Safety Study of the Inhibition of Agouti-related Protein (AgRP) for the Management of Obesity and Weight Loss
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: vTv Therapeutics (Industry)
Responsible Party: Jane Shen, Pharm.D., TransTech Pharma
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TTP435-201
Record Dates: First submitted 2008-10-23; First posted 2008-10-24 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2011-06

CONDITIONS: Obesity
Keywords: Obesity; Class 1; Class 2; Weight Loss; AgRP; TTP435; alphaMSH; Agouti-Related Protein; alpha-melanocyte stimulating hormone
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- TTP435 (Experimental)
  Interventions: Drug: TTP435

INTERVENTIONS:
Drug: TTP435
  Arms: TTP435
Drug: Placebo
  Arms: Placebo

SUMMARY:
Multiple pathways including peripheral and central hormones and neurotransmitters are involved in the regulation of food intake and body weight. One of the most studied pathways involves the melanocortin receptor. Agouti-related protein (AgRP) and alpha-melanocyte stimulating hormone (alphaMSH)have been shown to play an integral role in food intake and body weight.

It is reasonable to speculate that if there is an imbalance of alphaMSH and AgRP exist in obese individuals and inhibiting the activity of AgRP may be of therapeutic benefit in treating obesity.

ELIGIBILITY:
Inclusion Criteria:

* Male or female volunteers, aged 18 to 65 years, inclusive.
* Subjects must be obese (class 1: BMI of 30.0 to 34.9 kg/m2 or class 2: BMI of 35 to 39.9 kg/m2 in non-Asians and BMI of 27.0 - 31.9 kg/m2 or 32.0 - 36.9 kg/m2 in Asians) at the Screening Visit.
* Female subjects must be postmenopausal (with amenorrhea for at least 2 years prior to scheduled dosing and confirmatory FSH test in the range of 23-116 IU/L) or surgically sterile (with physician or insurance documentation of bilateral tubal ligation at least 6 months prior to Screening Visit or of a hysterectomy and/or bilateral oophorectomy) and agree not to undergo in vitro fertilization during the study and for 6 months post treatment.

Exclusion Criteria:

* Type 1 diabetes.
* Type 2 diabetes.
* History of myocardial infarction, stroke, including transient ischemic attack, in the last 2 years.
* Asthma or chronic obstructive pulmonary disease controlled by regular use of inhaled steroids.
* Subjects with rheumatoid arthritis, lupus, or multiple sclerosis regularly requiring steroids or disease-modifying anti-rheumatic agents.
* Subjects with psoriasis requiring oral steroids.
* Subjects planning to undergo gastric bypass or resection surgery, or who have had such a procedure in the 6 months prior to the Screening Visit.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2009-02; Primary Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Participant Adverse Events | Day 1 to Day 70 (2 weeks post dose)

SECONDARY OUTCOMES:
Change from Baseline Glucose Levels | Day 1 to Day 70 (2 weeks post dose)
Absolute Change in Body Weight | Day 1 to Day 70 (2 weeks post dose)
Absolute Change in Body Mass Index | Day 1 to Day 70 (2 weeks post dose)
Percent Change in Body Weight After 8 Weeks of Treatment with TTP435 or Placebo | Day 1 to Day 70 (2 weeks post dose)
Effect Subject-reported Satiety | Day 1 to Day 70 (2 weeks post dose)
Change from Baseline Insulin Levels | Day 1 to Day 70 (2 weeks post dose)
Change from Baseline Free Fatty Acid Levels | Day 1 to Day 70 (2 weeks post dose)
Change from Baseline Leptin Levels | Day 1 to Day 70 (2 weeks post dose)

CONTACTS AND LOCATIONS:
Overall Officials: James Wamsley, MD, Study Chair — vTv Therapeutics
Locations (12):
- United States (9):
  - Los Angeles, California
  - San Diego, California
  - Augusta, Georgia
  - Springfield, Illinois
  - Reno, Nevada
  - New York, New York
  - Charlotte, North Carolina
  - Norfolk, Virginia
  - Richmond, Virginia
- Canada (3):
  - Halifax, Nova Scotia
  - Oakville, Ontario
  - Toronto, Ontario